CLINICAL TRIAL: NCT05344846
Title: The Effect of Guided Imagery on Bonding and Breastfeeding After Cesarean; A Randomized Controlled Study
Brief Title: The Effect of Guided Imagery on Bonding and Breastfeeding After Cesarean
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Menekşe Nazlı AKER (Other)
Responsible Party: Sponsor-Investigator, Menekşe Nazlı AKER, Assist. Prof., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0555
Record Dates: First submitted 2022-04-19; First posted 2022-04-25 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Breastfeeding
MeSH Terms: conditions — Breast Feeding | interventions — Imagery, Psychotherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Guided imagery Group (Experimental): Guided imagery after cesarean
  Interventions: Other: Guided imagery
- Standard care (No Intervention): The participants in the control group will perform routine care of the clinic.

INTERVENTIONS:
Other: Guided imagery — The individuals in this group will be provided with guided imagery application. Guided imagery will be applied to the participants in the hospital environment 6-10 hours after the cesarean section. Afterwards, guided imagery application will be requested every day for two weeks.
  Arms: Guided imagery Group

SUMMARY:
The aim of this study is to evaluate the effect of guided imagery after cesarean section on mother-infant bonding and breastfeeding.

The study will be carried out in two different groups. The practice will start with meeting the women 6-10 hours after cesarean section. After the women are evaluated in terms of eligibility criteria for the research, the women who are eligible will be informed about the research and written informed consent will be obtained from the women who accept. The random distribution of women to the study groups will be carried out using the Block Randomization method. The following applications will be made to the groups.

Intervention Group; The individuals in this group will be provided with guided imagery application. Guided imagery will be applied to the participants in the hospital environment 6-10 hours after the cesarean section. Afterwards, guided imagery application will be requested every day for two weeks.

Control Group; The participants in the control group will perform routine care of the clinic.

ELIGIBILITY:
Inclusion Criteria:

* Nullipar
* Single birth
* Baby being with mother
* Gestational age 37-42 weeks
* Birth weight between 2500-4000 g
* APGAR score of 7 or higher in the 1st and 5th minutes
* The mother does not have a health problem that prevents breastfeeding
* Absence of conditions that prevent sucking, such as frenulum or palate problems

Exclusion Criteria:

* Participant's non-compliance with the research plan
* Interruption of breastfeeding for reasons such as health problems of the mother or baby
* Participants receive professional support for breastfeeding during the study process
* Hearing loss and deafness

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-05 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in how to feed baby | Baseline, 7th day, 14th day
  Nutrient content that she feeds her baby (Breastmilk, formula etc)
Change in The Mother-to-Infant Bonding Scale | Baseline, 7th day, 14th day
  The scale consists of eight adjectives (loving, resentful, neutral or felt nothing, joyful, dislike, protective, disappointed and aggressive), each followed by a four-point Likert scale ranging from "Very much" (0) to "Not at all" (5). When the adjective reflects a negative emotional response, the scoring is reversed. Thus, possible scores on the scale range between 0 and 24, with high scores indicating a problematic mother-to-infant bond (Taylor et al. 2005).
Change in Breastfeeding Self-Efficacy Scale | Baseline, 7th day, 14th day
  The 14-item scale was developed by Dennis (2003). The scale is a 5-point Likert-type scale (1= 'I am not sure at all' and 5 = 'I am always sure'). The scale's minimum score is 14 and the maximum score is 70. An elevated score shows an increase in breastfeeding self-efficacy.

SECONDARY OUTCOMES:
Change in Perception of Insufficient Milk Questionnaire | Baseline, 7th day, 14th day
  This scale, developed by McCarter-Spaulding for determining the perception of insufficient breast milk, is a six-question form. The scale's minimum score is 0 and the maximum score is 50. A high total score indicates that milk sufficiency perception is also high.

IPD SHARING:
Plan to Share IPD: Undecided